CLINICAL TRIAL: NCT04496479
Title: A Phase 2a, Open Label, Dose Escalation Study for Safety, Tolerability, and Efficacy of Hepatocyte Transplantation Into Periduodenal Lymph Nodes Among Subjects With End-Stage Liver Disease
Brief Title: Allogenic Hepatocyte Transplantation Into Periduodenal Lymph Nodes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LyGenesis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LYG-LIV-02-01
Record Dates: First submitted 2020-07-22; First posted 2020-08-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: End Stage Liver Disease
Keywords: Allogeneic; Organogenesis; Hepatocyte; Transplantation; Liver Disease
MeSH Terms: conditions — End Stage Liver Disease; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Open-Label Dose Escalation of Three Increasing Dosages
Masking Description: This is no masking in the open-label dose escalation phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LYG-LIV0001 (Experimental): Open label group of subjects with end stage liver disease receiving increasing doses of the experimental therapy.
  Interventions: Biological: LYG-LIV0001

INTERVENTIONS:
Biological: LYG-LIV0001 — Allogenic hepatocytes suspended in a buffered cell preservation solution with increasing number of lymph nodes being transplanted for the dose escalation. Subjects will also receive immune suppression, including tacrolimus capsules to follow the dose prescribed by the investigator as well as a short course of prednisone.

SUMMARY:
This Phase 2a clinical trial is a dose escalation study of the safety, tolerability, and efficacy of hepatocyte transplantation into lymph nodes via endoscopic ultrasound among subjects with end-stage liver disease.

DETAILED DESCRIPTION:
This safety, tolerability, and efficacy study includes an open-label dose-escalation phase for up to 12 subjects with end-stage liver disease (ESLD).

ELIGIBILITY:
Inclusion Criteria:

1. Have read, understood, and signed the informed consent form (ICF).
2. Adults of either gender and ages 18 to 70 years old with a diagnosis of ESLD due to alcohol, chronic hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infections, autoimmune hepatitis, primary sclerosis cholangitis, primary biliary cirrhosis (cholangitis), cirrhosis as the result of Wilson disease, hemochromatosis, sarcoidosis and alpha 1 antitrypsin deficiency, cryptogenic cirrhosis, and nonalcoholic steatohepatitis cirrhosis with a MELD-Na score >10 and <25 at screening.
3. Subjects must have a body mass index (BMI) <35.
4. Subjects with HCV associated ESLD must have been treated and demonstrate 24 weeks of negative HCV ribonucleic acid (RNA).
5. Subjects with HBV must be on stable therapy for 6 months and have HBV deoxyribonucleic acid <500 c/mL.
6. Women of childbearing potential (WOCBP) or sexual partners of male subjects who are WOCBP must be able and willing to use at least 1 highly effective method of contraception during the study and for 1 month after the last study visit. A female subject is considered to be a WOCBP after menarche and until she is in a postmenopausal state for 12 months or otherwise permanently sterile (for which acceptable methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy; HMA, 2014). For the definition and list of highly effective methods of contraception, see Appendix 1.
7. Has stable control of portal hypertension and upper gastrointestinal bleeding with medical therapy and/or endoscopic therapy.
8. If the subject has undergone a TIPS procedure for the clinical management of portal hypertension, they must be stable after the successful TIPS procedure, and not experiencing serious complications from the TIPS procedure itself (e.g., infection and intractable hepatic encephalopathy).
9. Has blood urea nitrogen (BUN) <80 mg/dL.
10. Has an estimated glomerular filtration rate (eGFR) ≥45 mL/min/1.73 m2.
11. Agrees to avoid alcohol consumption during the study.
12. Is willing and able to comply with all requirements of the study protocol.

Exclusion Criteria:

1. Has primary hepatic neoplasms (hepatocellular carcinoma and cholangiocarcinoma).
2. Has active and/or uncontrolled severe infections requiring hospitalization and prolonged antimicrobial therapy.
3. Has severe coagulopathy (international normalized ratio [INR] >2, and/or platelet count <50,000/μL).
4. Has psychiatric and/or social issues that could lead to noncompliance.
5. Has an extrahepatic neoplastic disease requiring active chemotherapy, immunotherapy, and/or surgical resection.
6. Has previously treated neoplastic disease with less than a 2-year cancer free period.
7. Pregnant and lactating women should not be in the study.
8. Known hypersensitivity to human serum albumin.
9. Subjects with uncontrolled hypertension (defined as a diastolic blood pressure of 110 mmHg or higher).
10. Has recurrent/intractable ascites refractory to diuretics and requiring periodic large volume paracentesis.
11. Has primary alcoholic liver disease and has not demonstrated abstinence for at least 24 weeks (6 months) prior to enrollment while attending mandatory rehab programs (e.g., Alcoholics Anonymous) and psychotherapy.
12. Has grade 3 esophageal varices requiring the continuous use of propranolol and cannot afford to have this medication withheld and/or discontinued.
13. Has a Child-Turcotte-Pugh (CTP) Class of C.
14. Is receiving or plans to receive treatment with another investigational product or device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Dosage Selection | Week 12
  The primary objective of the dose escalation is to confirm the optimal dose of transplanted hepatocytes to safely achieve adequate allogeneic hepatocyte (AH) engraftment
Safety of Engraftment of Hepatocytes in to Lymph Nodes | Week 12
  The primary safety objective of the dose escalation is to determine whether AH engraftments into the periduodenal lymph nodes in subjects with end-stage liver disease is safe as determined by the number/severity of adverse events
Efficacy of Engraftment of Hepatocytes in to Lymph Nodes | Week 12
  The primary efficacy objective of the dose escalation is to determine whether AH engraftments into the periduodenal lymph nodes in subjects with end-stage liver disease is efficacious in addressing some of the signs and symptoms of end-stage liver disease

SECONDARY OUTCOMES:
Effectiveness of Selected Treatment to Modify the Liver Function Panel | Week 52
  Evaluate the effectiveness of hepatocyte transplants in modifying the liver function panel (total serum bilirubin, ammonia, prothrombin time, international normalized ratio, sodium, blood urea nitrogen, and creatinine) as measured through changes in laboratory biomarkers caused by end-stage liver disease

OTHER OUTCOMES:
Change from Baseline in Ascities/Sarcopenia | Week 52
  Changes from baseline in ascities/sarcopenia as measured by Computerized Tomography (CT) Scan
Change from Baseline in Lean Body Mass | Week 52
  Changes from baseline in lean body mass as measured by Skinfold Testing, Bioelectrical Impedance Analysis, or DexaScan
Change from Baseline in Liver Reserve | Week 52
  Changes from baseline in liver reserve as measured through the Disease Severity Index
Change from Baseline in Hepatic Function | Week 52
  Changes from baseline in hepatic function as measured through the HepQuant SHUNT Testing (assessing liver function in chronic liver disease)
Change from Baseline in Quality of Life | Week 52
  Changes from baseline in quality of life as measured through the SF-36 (total score and sub-scale scores) Questionnaire
Change from Baseline in Fatigue | Week 52
  Changes from baseline in fatigue as measured through the Neuro-QOL Short Form (Fatigue Scale)
Change from Baseline in Neuropsychological Status | Week 52
  Changes from baseline in neuropsychological status as measured by the Repeatable Battery of Neuropsychological Status (RBANS) test

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Fontes, MD, Study Chair — LyGenesis, Inc.
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No